CLINICAL TRIAL: NCT00339950
Title: Diet, Other Risk Factors, Genetics and the Risk of Colorectal Neoplasia in a Screening Trial of Asymptomatic Women: A Sub-Study of the CONCeRN Trial
Brief Title: Colorectal Neoplasia Screening w Colonoscopy in Asymptomatic Women at Regional Navy/Army Medical Ctrs: The CONCeRN Trial
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999900010; OH00-C-N010
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Adenoma
Keywords: Colorectal adenoma; Screening; Diet; Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood, colon tissue

GROUPS / COHORTS (1):
- 1: Asymptomatic women between the ages of 40 and 75 referred to regional military medical centers for routine colorectal screening

SUMMARY:
The CONCeRN Trial is a multi-center study of asymptomatic women between the ages of 40 and 75 referred to regional military medical centers for routine colorectal screening. The primary purpose of the main study is to determine the extent to which advanced neoplastic lesions will be missed if clinicians only perform sigmoidoscopies rather than full colonoscopies as a screening procedure and to resolve current debate about the significance of sigmoidoscopic detection of single, small, tubular adenomas (i.e., do they imply greater risk for large adenomatous polyps or colorectal cancer at other sites beyond the reach of the sigmoidoscope, or is there no increased risk?). Women enrolled in the trial receive colonoscopy during which all identified polyps are removed and also during which two pinch biopsies of apparently-normal tissue are taken. In addition, before the colonoscopy is performed, patients wil have blood drawn and answer a brief questionnaire on risk factors for colorectal cancer. The sub-study proposes to add on a more extensive questionnaire to assess dietary and other lifesyle factors potentially related to colorectal cancer, and to draw additional blood for assessment of nutritional status and for analysis of genetic polymorphisms related to colorectal cancer. With the additional information available from these questionnaires and blood samples, it will be possible to explore the extent to which various dietary and genetic risk factors are related to colorectal polyps in asymptomatic women of average risk for disease.

DETAILED DESCRIPTION:
The CONCeRN Trial is a multi-center study of asymptomatic women between the ages of 40 and 75 referred to regional military medical centers for routine colorectal screening. The primary purpose of the main study is to determine the extent to which advanced neoplastic lesions will be missed if clinicians only perform sigmoidoscopies rather than full colonoscopies as a screening procedure and to resolve current debate about the significance of sigmoidoscopic detection of single, small, tubular adenomas (i.e., do they imply greater risk for large adenomatous polyps or colorectal cancer at other sites beyond the reach of the sigmoidoscope, or is there no increased risk?). Women enrolled in the trial receive colonoscopy during which all identified polyps are removed and also during which two pinch biopsies of apparently-normal tissue are taken. In addition, before the colonoscopy is performed, patients will have blood drawn and answer a brief questionnaire on risk factors for colorectal cancer. The NCI-led sub-study added a more extensive questionnaire to assess dietary and other lifestyle factors potentially related to colorectal cancer, and obtained additional blood for assessment of nutritional status and for analysis of genetic polymorphisms related to colorectal cancer. With the additional information available from these questionnaires and blood samples, it will be possible to explore the extent to which various dietary and genetic risk factors are related to colorectal polyps in asymptomatic women of average risk for disease. Recruitment is now complete at all sites. A total of 937 women were recruited. Of these, about one-quarter of the women with one or more adenomas had an advanced adenoma, defined as being greater than or equal to 1 cm in diameter, or having high grade dysplasia or villous elements). These neoplasia prevalence figures are in line with initial projections. Active contact with participants is concluded. We have now entered into a data analysis phase.

ELIGIBILITY:
* INCLUSION CRITERIA:

50-79, asymptomatic women of average risk referred for colorectal screening.

40-79 year-old asymptomatic women referred for colorectal screening with a history of colorectal cancer in a first degree relative.

EXCLUSION CRITERIA:

History of positive stool guiaic within six months of referral.

History of iron deficiency anemia within six months of referral (Note: if patients have not had stool guiacs, complete blood cell count or ferritin performed within the last six months, then these tests will be performed at time of study enrollment).

History of normal colonoscopy or barium enema within past ten years or history of normal flexible sigmoidoscopy within past 5 years.

History of adenomatous polyps, colorectal cancer, inflammatory bowel disease, HNPCC, or familial adenomatous polyposis.

History of rectal bleeding or hematochezia within the past 12 months.

Unintentional weight loss greater than 10 pounds within previous six months.

Pregnant women.

Subjects under 18 years of age.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic women between the ages of 40 and 75 referred to regional military medical centers for routine colorectal screening@@@
Sampling Method: Non-Probability Sample
Enrollment: 937 (Actual)
Dates: Start 2000-02-14 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Sinha, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Naval Medical Center, San Diego, San Diego, California
  - National Naval Medical Center, Bethesda, Maryland
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia

REFERENCES:
- [Background] Adamson RH, Thorgeirsson UP, Snyderwine EG, Thorgeirsson SS, Reeves J, Dalgard DW, Takayama S, Sugimura T. Carcinogenicity of 2-amino-3-methylimidazo[4,5-f]quinoline in nonhuman primates: induction of tumors in three macaques. Jpn J Cancer Res. 1990 Jan;81(1):10-4. doi: 10.1111/j.1349-7006.1990.tb02500.x. PMID 1691162
- [Background] Bosron WF, Li TK. Genetic polymorphism of human liver alcohol and aldehyde dehydrogenases, and their relationship to alcohol metabolism and alcoholism. Hepatology. 1986 May-Jun;6(3):502-10. doi: 10.1002/hep.1840060330. PMID 3519419
- [Background] Boutron MC, Faivre J, Marteau P, Couillault C, Senesse P, Quipourt V. Calcium, phosphorus, vitamin D, dairy products and colorectal carcinogenesis: a French case--control study. Br J Cancer. 1996 Jul;74(1):145-51. doi: 10.1038/bjc.1996.330. PMID 8679449